CLINICAL TRIAL: NCT01261026
Title: Are Serum Levels of Vascular Endothelial Growth Factor a Marker for the Early Diagnosis of Ectopic Pregnancy?
Acronym: UNIFESP
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Other Study IDs: JEJ-060866
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2007-12

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Ectopic pregnancy, extra-uterine pregnancy: Ectopic pregnancy, control
- Abnormal intrauterine pregnancy

SUMMARY:
OBJECTIVE: This study evaluated serum vascular endothelial growth factor (VEGF) concentrations in women with ectopic pregnancy (EP), abnormal intrauterine pregnancy (aIUP) and normal intrauterine pregnancy (nIUP).

METHODS: This was a prospective, case-control study comparing serum VEGF concentrations among 72 women with ectopic pregnancy (n=35), abnormal IUP (n=15) and normal IUP (n=22) matched for gestational age. For the determination of serum VEGF concentration a solid phase sandwich ELISA was used. Patients were stratified according to serum VEGF above or below 200pg/mL.

RESULTS: The serum level of VEGF was significantly higher in women with ectopic pregnancy (median 211.1 pg/mL; range 5 - 1017.0 pg/mL) than in women with normal IUP (median 5 pg/mL; range 5- 310.6 pg/mL) P < 0.0001. Serum VEGF concentrations did not show any statistically significant difference between women with aIUP (median 231.9 pg/mL range 5 - 813.7 pg /mL ) and EP (median 211.1 pg/mL range 5 - 1017.0 pg/mL). When cut-off concentrations of 200 pg/mL for VEGF were used, a nIUP could be distinguished from an unviable (EP and aIUP) with a sensitive of 53%, specificity of 90.9%, a positive predictive value of 92.9% and a negative predictive value of 46.5%..

CONCLUSIONS: Serum VEGF could not distinguish between an EP and an aIUP. However, serum VEGF concentrations above 200 pg/mL could discriminate a nIUP from an unviable pregnancy (EP or aIUP) with a PPV of 92.9%.

ELIGIBILITY:
Inclusion Criteria:The inclusion criterion was the presence at transvaginal ultrasound of an extraovarian adnexal mass in women with a suspected ectopic pregnancy (amenorrhea, bleeding and pain) with positive test for beta-hCG.

-

Exclusion Criteria:The exclusion criterion was non-tubal ectopic pregnancy (cervical, cesarean scar, ovarian, and abdominal).

-

Ages: 15 Years to 40 Years | Sex: Female
Age Groups: Child, Adult
Study Population: ectopic pregnancy abnormal intrauterine pregnancy normal intrauterine pregnancy
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Ugurlu EN, Ozaksit G, Karaer A, Zulfikaroglu E, Atalay A, Ugur M. The value of vascular endothelial growth factor, pregnancy-associated plasma protein-A, and progesterone for early differentiation of ectopic pregnancies, normal intrauterine pregnancies, and spontaneous miscarriages. Fertil Steril. 2009 May;91(5):1657-61. doi: 10.1016/j.fertnstert.2008.02.002. Epub 2008 Apr 9. PMID 18402945
- [Result] Daponte A, Pournaras S, Zintzaras E, Kallitsaris A, Lialios G, Maniatis AN, Messinis IE. The value of a single combined measurement of VEGF, glycodelin, progesterone, PAPP-A, HPL and LIF for differentiating between ectopic and abnormal intrauterine pregnancy. Hum Reprod. 2005 Nov;20(11):3163-6. doi: 10.1093/humrep/dei218. Epub 2005 Jul 29. PMID 16055453